CLINICAL TRIAL: NCT03622697
Title: Mindfulness Meditation to Improve Social Functioning and Quality of Life in Patients With Facial Paralysis: A Randomized Controlled Trial
Brief Title: Effects of Mindfulness Meditation on Facial Paralysis Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study expired in IRB.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00135870
Record Dates: First submitted 2018-08-03; First posted 2018-08-09 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-06

CONDITIONS: Facial Paralysis
Keywords: mindfulness; meditation; facial paralysis; quality of life; social functioning
MeSH Terms: conditions — Facial Paralysis; Social Adjustment

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Meditation Arm (Experimental): Mindfulness meditation intervention: patients will be asked to complete a guided mindfulness meditation phone application intervention.
  Interventions: Behavioral: Mindfulness Meditation Phone Application
- Non-Intervention Arm (No Intervention): Patients assigned to the non-intervention arm will not be instructed to use a mindfulness meditation phone application and instead will listen to educational materials.

INTERVENTIONS:
Behavioral: Mindfulness Meditation Phone Application — Mindfulness meditation intervention: patients will be asked to complete a guided mindfulness meditation intervention using a phone application for at least 4 weeks with periodic survey assessments using validated psychometric tools.
  Arms: Mindfulness Meditation Arm

SUMMARY:
Currently, physicians have several options in addressing the anatomic and physiologic sequela of facial paralysis. However, strategies to address the psychologic and coping ability for patients have not been investigated.

The goal is to investigate the effect of mindfulness meditation on social functioning in patients with facial paralysis. This study will also explore whether increasing social functioning in patients with facial paralysis will improve overall quality of life. These questions will be answered using a randomized controlled trial.

DETAILED DESCRIPTION:
In this study population, facial paralysis was significantly associated with increased loneliness, decreased social function, decreased comfort with socializing, and worse quality of life scores. Furthermore, prior studies have shown that facial paralysis increases the likelihood of depression as measured on validated psychometric instruments. Currently, treating physicians have several options in addressing the anatomic and physiologic sequela of facial paralysis. However, strategies to address the psychologic and coping ability for patients have not been investigated. To better provide patient-centered care, physicians should consider the psychosocial impact of facial paralysis to identify patients who may benefit from additional support interventions to complement facial reanimation treatment plans.

This is a prospective repeated measures study examining psychosocial status as measured by validated psychometric instruments. The intervention group will participate in mindfulness meditation using a phone application. Assessment of social functioning and quality of life will be conducted using survey instruments.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age
* Must have any-cause facial paralysis

Exclusion Criteria:

* Patients younger than 18 years old
* Non-English speakers
* Patients without smart-phone access
* Patients with autism
* Patients with schizophrenia
* Patients with an affective psychiatric condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Social Functioning as assessed by University of California, Los Angeles 3-point loneliness scale | Change from baseline at 2 weeks, 4 weeks, and 6 weeks
  University of California, Los Angeles 3-point loneliness scale - minimum score 0, maximum score 100 assessing how often one feels socially isolated, higher indicating greater loneliness
Changes in Social Functioning as assessed by Facial Disability Index | Change from baseline at 2 weeks, 4 weeks, and 6 weeks
  Facial disability index (social functioning portion) - categorical responses ranging from "never" to "all of the time" for social problems associated with facial muscle function over the past month to measure social functioning; the minimum to maximum score range for social functioning is 5 to 30 with a higher score indicating greater social functioning
Changes in Social Functioning as assessed by a Social Functioning Visual Analog Scale | Change from baseline at 2 weeks, 4 weeks, and 6 weeks
  Social functioning visual analog scale - single-item questionnaire ranging from 0 to 100 with greater numbers indicating more comfort in socializing with others

SECONDARY OUTCOMES:
Changes in Reported Quality of Life as assessed by a Visual Analog Scale | Change from baseline at 2 weeks, 4 weeks, and 6 weeks
  Quality of life will be measured using the validated quality of life visual analog scale (single-item questionnaire ranging from 0 to 100 with greater numbers indicating a higher quality of life)
Changes in Anxiety assessed by the State-Trait Anxiety Inventory | Change from baseline at 2 weeks, 4 weeks, 6 weeks
  Anxiety will be measured using the validated State-Trait Anxiety Inventory with 20 items measuring trait anxiety and 20 items measuring state anxiety, each with categorical responses ranging from "never" to "very much so" in response statements regarding how one feels generally (trait) and at the current moment (state)
Changes in Mindfulness as measured using the Cognitive and Affective Mindfulness Scale-Revised | Change from baseline at 2 weeks, 4 weeks, 6 weeks
  Mindfulness will be measured using the validated Cognitive and Affective Mindfulness Scale-Revised which is a 12-item questionnaire with categorical responses ranging "rarely/not at all" to "almost always" regarding statements about one's experience of mindfulness with minimum score of 12 points to a maximum score of 48 points where a higher score indicates greater mindful qualities
Changes in Physical Functioning as assessed by Facial Disability Index | Change from baseline at 2 weeks, 4 weeks, 6 weeks
  Facial disability index (physical functioning portion) - categorical responses ranging from "usually with no difficulty" to "usually did not do because of health" for physical problems associated with facial muscle function over the past month to measure physical functioning; the minimum to maximum score range for social functioning is 0 to 25 with a higher score indicating worse physical function

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Ishii, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Johns Hopkins - Green Spring Station, Lutherville-Timonium, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoge EA, Bui E, Palitz SA, Schwarz NR, Owens ME, Johnston JM, Pollack MH, Simon NM. The effect of mindfulness meditation training on biological acute stress responses in generalized anxiety disorder. Psychiatry Res. 2018 Apr;262:328-332. doi: 10.1016/j.psychres.2017.01.006. Epub 2017 Jan 26. PMID 28131433
- [Background] Simkin DR, Black NB. Meditation and mindfulness in clinical practice. Child Adolesc Psychiatr Clin N Am. 2014 Jul;23(3):487-534. doi: 10.1016/j.chc.2014.03.002. PMID 24975623
- [Background] Nellis JC, Ishii M, Byrne PJ, Boahene KDO, Dey JK, Ishii LE. Association Among Facial Paralysis, Depression, and Quality of Life in Facial Plastic Surgery Patients. JAMA Facial Plast Surg. 2017 May 1;19(3):190-196. doi: 10.1001/jamafacial.2016.1462. PMID 27930763